CLINICAL TRIAL: NCT05284565
Title: Concordance Between the Electromedical Device Nexkin DSPT and the Manual Procedure in the Measurement of Papules in Allergy Skin Testing
Brief Title: Comparative Study of Skin Prick Allergy Test Measurements Between Current Manual Procedure and Nexkin DSPT Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: INNOPRICK SL (Industry)
Collaborators: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NEXKIN01
Record Dates: First submitted 2022-02-25; First posted 2022-03-17 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Allergy
Keywords: skin prick test; allergy; skin testing; SPT; 3D imaging; allergy testing; allergy test reading; automatic measurement
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: The study will prospectively include patients attending the Allergology Department, after signing an informed consent form and a data protection clause.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Results of reading (Other): All patients who were prick tested and accepted to participate in the study, were prospectively included in the study in only one arm. All of their tests were read by the device and the manual procedure.
  Interventions: Device: Reading of the skin prick allergy test

INTERVENTIONS:
Device: Reading of the skin prick allergy test — A double reading of the forearm will be performed with the Nexkin DSPT device. Also, two healthcare professionals will perform, consecutively, the manual reading according to their usual practice. Nexkin DSPT device provides a semi-automatic wheal detection, presenting the user an initial set of potential wheals and information about them (as their measure).
  Healthcare professional can then discard, add and/or confirm wheals by visual validation, and add/edit wheal information. The device automates the test reading process, digitises the results, and quantifies.

SUMMARY:
Clinical trial with the aim to evaluate the level of agreement in wheal size measures in allergy skin prick testing (SPT) between the electro-medical device Nexkin DSPT® and the manual measurement procedure used in the daily practice.

DETAILED DESCRIPTION:
The purpose of the trial is to evaluate the concordance of measurements obtained by the Nexkin DSPT device versus the measurements obtained manually.

A prospective clinical trial study was conducted at Clínica Universidad de Navarra. SPT will be tested in the same way as during a routine visit, with the only difference being that the images of the arm required for the device to operate will be captured. Nexkin DSPT device is a non-invasive device, which does not perform the procedure of puncture and appearance of papules. The device is only used to read the test results. There is no risk to the patient or the healthcare professionals involved in capturing images with the device. Device does not provide a diagnosis and it is not a substitute for sound medical judgment.

The study will prospectively include patients attending the allergy consultation (sample size calculated in 93 patients) with positive (histamine) and negative (saline solution) controls. Fifteen minutes later, two consecutive readings with the device and two manual readings were performed by two different nurses. The area of the histamine wheals was measured automatically by Nexkin DSPT and after the manual procedure measured manually by planimetry.

ELIGIBILITY:
Inclusion Criteria:

1. Patient to be tested with aeroallergen and/or food battery prick tests.
2. Patient over 12 years of age.
3. Patient, or his/her representative, who has given consent to participate in the study.
4. Patient who has not taken an antihistamine for more than 3 days.
5. Women of childbearing age who, at the time of taking the clinical history, declare that they are not pregnant.

Exclusion Criteria:

1. Patients who are to be tested with a prick number greater than 40.
2. Patients who are to be tested with a prick number less than 40, but for whom it is necessary to place more than two rows of allergens in at least one of the arms.
3. Patients who have taken an antihistamine within the previous 3 days.
4. Patients who are being treated with antidepressants or other drugs with an antihistamine effect.
5. Patients who suffer severe atopic dermatitis affecting the forearms.
6. Patients with dermographism.
7. Patients who are to undergo intradermal testing.
8. Pregnant women or women suspected of pregnancy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Agreement in wheal size measures in allergy skin testing between the electro-medical device Nexkin DSPT and the manual measurement procedure | 5 minutes
  Fifteen minutes after the punctures have been performed, a double reading of the forearm shall be taken with the device. The first reading will be stored for later analysis, and the second reading will be used afterwards. The healthcare professional will then perform the manual reading and generate the manual result sheet as is standard practice.
  The health professional visually examines the forearm and compares his observation with the identification presented by the device.
  The result of the identifications made by the device as well as the interactions of the healthcare professional on the screen shall be recorded on the device.
  Diameter measurements are measured in millimetres (mm) and area measurements are measured in square millimetres (mm2).

SECONDARY OUTCOMES:
Test-retest reliability of device reading. | 5 minutes
  15 minutes after the punctures have been performed, a double reading of the forearm shall be taken with the device. The first reading will be stored for later analysis, and the second reading will be used afterwards. The healthcare professional will then perform the manual reading and generate the manual result sheet as is standard practice.
  The health professional visually examines the forearm and compares his observation with the identification presented by the device.
  The result of the identifications made by the device as well as the interactions of the healthcare professional on the screen shall be recorded on the device.
  Diameter measurements are measured in millimetres (mm) and area measurements are measured in square millimetres (mm2).
Variability in measurements of histamine wheals made by different health professionals. | 5 minutes
  15 minutes after the punctures have been performed, a reading of the forearm will be performed by the device. Then, a first healthcare professional will perform the manual reading and generate the manual result sheet as in standard practice.
  Immediately afterwards, the first professional will erase the contours of the wheals on the forearm of the patient. A second healthcare professional will perform the manual reading without knowing the reading performed by the first one, and will generate the manual result sheet as is done in routine practice.
  The reading order of each test between the two healthcare professionals is randomised.
  Diameter measurements are measured in millimetres (mm) and area measurements are measured in square millimetres (mm2).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Gastaminza Lasarte, Dr., Principal Investigator — Clinica Universidad de Navarra, Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Universidad de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Justo X, Diaz I, Gil JJ, Gastaminza G. Medical Device for Automated Prick Test Reading. IEEE J Biomed Health Inform. 2018 May;22(3):895-903. doi: 10.1109/JBHI.2017.2680840. Epub 2017 Mar 9. PMID 28362597
- [Background] Justo X, Diaz I, Gil JJ, Gastaminza G. Prick test: evolution towards automated reading. Allergy. 2016 Aug;71(8):1095-102. doi: 10.1111/all.12921. Epub 2016 May 20. PMID 27100940
- [Background] Morales-Palacios MP, Nunez-Cordoba JM, Tejero E, Matellanes O, Quan PL, Carvallo A, Sanchez-Fernandez S, Urtasun M, Larrea C, Iniguez MT, Gimenez R, Goikoetxea MJ, D'Amelio CM, Ferrer M, Gastaminza G. Reliability of a novel electro-medical device for wheal size measurement in allergy skin testing: An exploratory clinical trial. Allergy. 2023 Jan;78(1):299-301. doi: 10.1111/all.15474. Epub 2022 Aug 20. No abstract available. PMID 35950712